CLINICAL TRIAL: NCT06866457
Title: Effectiveness of an Audio-hypnosis Intervention on Pre-interventional Anxiety During an MRI Examination in Children and Adolescents: a Randomized Controlled Trial
Brief Title: Audio Hypnosis for Reducing Anxiety in Children and Adolescents Undergoing MRI: A Randomized Controlled Trial
Acronym: EKHyp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 260/2024
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hypnosis; Anxiety, Preoperative
Keywords: MRI Anxiety in Children; Hypnosis in Pediatric Medicine; hypnosis; hypnosis MRI
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: the MRI technologists are blinded outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypnosis group (Experimental): listen to an audio hypnosis via a digital recording ("Elli's dream story"), which is accessible via a QR code, before the MRI examination
  Interventions: Other: Audio hypnosis
- Control group (No Intervention): Standard pre-MRI information provided by medical staff

INTERVENTIONS:
Other: Audio hypnosis — Audio hypnosis via a digital recording ("Ellis Traumgeschichte") accessible via QR code
  Arms: hypnosis group

SUMMARY:
The goal of this clinical trial is to find out if listening to an audio hypnosis recording can help reduce anxiety in children and adolescents (ages 6-14) who are getting an MRI scan without sedation. The main questions the study will answer are:

Does listening to a hypnosis audio before an MRI help children feel less anxious? Can hypnosis audio help reduce scan interruptions or early terminations?

To find out, researchers will compare one group of children who listen to the hypnosis audio with another group who receive the usual explanation from medical staff to see if the audio helps lower anxiety and makes the MRI process smoother.

What participants will do:

Be randomly placed into either the hypnosis group (who get access to the hypnosis audio) or the control group (who receive the usual explanation).

Listen to the hypnosis audio as many times as they like before the MRI (if in the hypnosis group).

Fill out questionnaires before and after the MRI to measure anxiety (both children and parents).

Have their MRI scan while researchers track any interruptions or early terminations.

Have their anxiety levels rated by MRI technologists after the scan.

This study aims to see if a simple, non-medication method like audio hypnosis can help children feel calmer during MRI exams.

DETAILED DESCRIPTION:
Study Overview This is a randomized controlled trial (RCT) investigating the effectiveness of an audio hypnosis intervention in reducing pre-procedural anxiety in children and adolescents (ages 6-14) undergoing an MRI examination without sedation. The study will compare an intervention group (receiving access to an audio hypnosis recording) with a control group (receiving standard pre-MRI explanations) to assess whether the hypnosis audio reduces anxiety levels, improves patient cooperation, and minimizes scan interruptions or movement artifacts.

The study is monocentric, conducted at the Elisabeth Hospital Essen, Department of Pediatric Medicine, and aims to enroll 100 participants (50 per group).

Study Design

* Type: Randomized, controlled, single-center interventional study
* Intervention: Audio hypnosis via a digital recording ("Ellis Traumgeschichte") accessible via QR code
* Control: Standard pre-MRI information provided by medical staff
* Sample Size: 100 participants (50 per group)
* Study Duration: Recruitment period of up to 24 months, with the total study duration extending until data analysis is complete
* Intervention Duration: The hypnosis audio lasts approximately 20 minutes and can be listened to multiple times before the MRI scan Intervention and Data Collection

Participants will be randomly assigned to one of two groups:

* Intervention Group: Receives a flyer with a QR code linking to a hypnosis audio recording, which they can listen to as often as they wish before their MRI scan.
* Control Group: Receives standard verbal and written pre-MRI information from medical staff without additional hypnosis intervention.
* Both Groups: Undergo their scheduled MRI scan and receive routine medical counseling.

Data Collection Time Points:

* T0 (Baseline):

  * Participant enrollment, informed consent, and randomization
  * Distribution of hypnosis audio (intervention group only)
* T1 (Before MRI):

  * Self-reported anxiety assessment using the KAT III questionnaire
  * Parent-reported anxiety assessment using a visual analog scale (VAS)
* T2 (During MRI):

  * Recording of scan interruptions
  * Noting if the MRI scan was terminated early
  * Presence of motion artifacts on MRI images
* T3 (After MRI):

  * Retrospective self-reported anxiety assessment using KAT III
  * MRI technologist's anxiety assessment using VAS Registry and Data Quality Assurance Measures

Although this study is not a formal patient registry, strict data quality control measures will be implemented to ensure the accuracy and reliability of collected data:

1. Quality Assurance Plan:

   * The study will adhere to Good Clinical Practice (GCP) guidelines, with regular monitoring and documentation audits.
   * Data validation checks will be applied to ensure consistency in reported anxiety levels across time points.
   * Any protocol deviations will be recorded and evaluated.
2. Data Validation and Range Checks:

   * Automated range checks will be implemented to detect inconsistencies in questionnaire responses (e.g., unrealistic changes in anxiety scores).
   * Manual verification of data entries will be performed by research staff.
3. Source Data Verification (SDV):

   * Randomly selected data entries will be compared with original records (e.g., consent forms, MRI technologist logs) to ensure accuracy.
   * Adherence to protocol-defined randomization procedures will be confirmed.
4. Data Dictionary:

   * Variables include demographic data, anxiety scores (KAT III, VAS), scan interruptions, and MRI completion rates.
   * Standardized coding and response scales (e.g., VAS range 0-10) will be used to maintain consistency across participants.
5. Standard Operating Procedures (SOPs):

   * Detailed SOPs will be followed for patient recruitment, randomization, intervention administration, data collection, and adverse event monitoring.
   * Adverse events, though unlikely, will be recorded and reported according to ethical guidelines.
6. Sample Size Assessment:

   * Based on literature data, a medium effect size (Cohen's d = 0.60) was assumed for pre-MRI anxiety reduction.
   * 90 participants (45 per group) are required to achieve 80% power at α = 0.05 using a two-sided t-test.
   * To account for a 10% dropout rate, 100 participants will be enrolled (50 per group).
7. Handling of Missing Data:

   * Missing questionnaire responses will be managed using multiple imputation techniques via the Markov Chain Monte Carlo (MCMC) method.
   * Sensitivity analyses will be performed to assess the impact of missing data on study conclusions.
8. Statistical Analysis Plan:

   * The primary hypothesis (anxiety reduction in the intervention group) will be tested using a two-sided t-test with a significance level of α = 0.05.
   * Secondary outcomes will be analyzed using linear mixed models to account for repeated measures.
   * The intention-to-treat (ITT) principle will be applied to all analyses.
   * The potential mediation effect of reduced anxiety on MRI scan success (fewer interruptions, better image quality) will be explored using regression models.

Risk and Benefit Assessment

* Potential Benefits:

  * Reduction of MRI-related anxiety in children without the need for sedation
  * Potential for fewer MRI scan interruptions and better image quality
  * Non-invasive, low-cost, and easily scalable intervention
* Potential Risks:

  * Minimal risks, comparable to standard relaxation techniques
  * Some participants may experience mild side effects (e.g., dizziness, headache) Ethical and Regulatory Considerations
* Ethical approval: The study was approved by the Ethics Committee of Witten/Herdecke University
* Informed Consent:

  * Participants and their parents will receive detailed study information and provide written informed consent.
  * Withdrawal from the study is possible at any time without consequences.
* Data Protection:

  * All study data will be pseudonymized to protect participant confidentiality.
  * Data will be stored in secure, access-controlled databases and used exclusively for research purposes.

Funding and Sponsorship

* The study is not externally funded.
* The development of the hypnosis intervention and study materials was supported by Ellis Freunde, a non-profit organization.
* No financial conflicts of interest exist for the study investigators. Conclusion This randomized controlled trial aims to provide scientific evidence on the effectiveness of audio hypnosis as a simple, non-pharmacological intervention to reduce MRI-related anxiety in children and adolescents. The study incorporates rigorous data quality assurance measures, follows GCP-compliant protocols, and implements a robust statistical analysis plan to ensure reliable and meaningful results.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 14 years
* Planned MRI examination without anesthesia
* Subjects should have a good understanding of the German language

Exclusion Criteria:

* Severe cognitive impairment or mental retardation
* Severely limiting psychiatric disorders
* Addictive disorders
* Limited understanding of the German language
* Taking sedative medication (e.g. lorazepam)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
anxiety prosective | directly before the MRI
  Self-reported anxiety assessment using the KAT III questionnaire

SECONDARY OUTCOMES:
Anxiety External assessment by parents | directly before the MRI
  Anxiety External assessment by parents (Visual Analog Scale (VAS)
MRI Interruption frequency, Cancellation, Motion artifacts | during MRI
  MRI Interruption frequency, Cancellation, Motion artifacts on MRI images by MRI technologists
Anxiety external assessment by MRI technologist | directly after MRI
  Anxiety external assessment by MRI technologist using VAS (visual analog scale)
Anxiety retrospective | directly after MRI
  Retrospective self-reported anxiety assessment using KAT III questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Elisabeth Hospital, Essen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
available upon request from Dr. med. Melanie Anheyer (m.anheyer@contilia.de)